CLINICAL TRIAL: NCT06055946
Title: Prospective, Multicenter, Single-arm Study on the Performance of Symmcora® Long-term Bidirectional Barbed Suture for Vesicourethral Anastomosis in Patients Undergoing Robot Assisted Radical Prostatectomy.
Brief Title: Symmcora® Long-term Bidirectional Barbed Suture for Anastomosis in Patients Undergoing Robot Assisted Radical Prostatectomy
Acronym: BARVANA LONG
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2207
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: robot assisted radical prostatectomy; barbed suture
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symmcora® Long bidirectional: Symmcora® Long-term bidirectional barbed suture for vesicourethral anastomosis in patients undergoing robotic assisted radical prostatectomy.
  Interventions: Device: robotic assisted radical prostatectomy

INTERVENTIONS:
Device: robotic assisted radical prostatectomy — Adult male patients undergoing elective robotic assisted radical prostatectomy.will be included in the study

SUMMARY:
The aim of this observational study is to show the superiority of the bidirectional barbed suture (Symmcora® Longterm) in terms of time to perform the vesicourethral anastomosis after robot assisted radical prostatectomy compared to the available literature data, without an increase in the complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Male patients undergoing an elective robotic assisted radical prostatectomy
* Written informed consent
* Age ≥ 18years

Exclusion Criteria:

* Emergency surgery
* History of chronic steroid use
* Previous prostatic surgery
* Previous radiotherapy or brachytherapy
* Patients with hypersensitivity or allergy to the suture material.
* Participation in another study
* Non-compliant patient (dementia etc)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients undergoing an elective robotic assisted radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Time to perform the vesicourethral anastomosis | intraoperatively
  Time to perform the vesicourethral anastomosis using a stopwatch. Time starts when the needle passes the first time the tissue and ends after completion of the anastomosis. Completion of the anastomosis is defined by the last cut of the thread.

SECONDARY OUTCOMES:
Anastomotic leak rate until 6 months postoperatively | up to 6 months after surgery
  Cumulative number of anastomotic leaks
Amount of estimate blood loss (EBL) | intraoperatively
  Blood loss is estimated by the amount of intraoperatively needed transfusion
Transfusion rate | at discharge from hospital (approximately 5-10 days after surgery)
  Amount of transfused blood, Calculated by multiplication of the number of bags needed and the volume in ml per bag
Urinary retention | at 6 weeks postoperatively
  Urinary retention is an inability to completely empty the bladder
Urinary fistula rate | until 6 months postoperatively
  A urogenital fistula is an abnormal tract that exists between the urinary tract and bladder, ureters, or urethra. A urogenital fistula can occur between any of the organs and structures of the pelvic region. A fistula allows urine to continually exit through and out the urogenital tract.
Bladder neck contracture rate | until 6 months postoperatively
  Cumulative rate of patients with a complication related to the bladder neck contracture
Urinary stone formation rate | until 6 months postoperatively
  Cumulative rate of patients with a complication related to urinary stone formation
Rate of other complications | until 6 months postoperatively
  Cumulative rate of patients with any other complication (infection, embolization, peritonitis, ileus, etc.)
Operation consola time | intraoperatively
  Time to perform the intervention from first cut to last cut of the last thread. The time is measured using a stopwatch.
Time to perform the Rocco stitch | intraoperatively
  Time to perform the modified Rocco stitch: After prostate extirpation, the free edge of the Denonvillier fascia is approximated to the posterior rhabdosphincter/median raphe using a running suture. Then, the Denonvilliers' fascia is fixated to the posterior wall of the bladder, which reduces tension in the anastomosis and provides pelvic support to the bladder neck. The time is measured using a stopwatch.
Length of postoperative stay | until discharge (approximately 5-10 days postoperatively)
  Number of days from surgery till patient is discharged from hospital
Catheterization duration | until first follow-up (6 weeks postoperatively)
  Number of days from surgery till catheter was finally removed
Early continence | 6 weeks postoperatively
  Days after catheter was finally removed to complete continence
Development of continence by 24-h pad test | at 3 months and 6 months postoperatively.
  The 24-hour pad test is used as an objective diagnostic method for the assessment of post prostatectomy stress urinary incontinence. Pads are weighed before and after use and the amount of urine is measured.
Development of Erectile Function compared to baseline | Preoperatively (Baseline), 6 weeks, 3 months and 6 months postoperatively.
  Erectile Function measured by International Index of Erectile Function (IIEF-5). The International Index of Erectile Function-5 (IIEF-5) is an five-item Index developed to diagnose the presence and severity of erectile dysfunction (ED). The five items are based on ability to identify the presence or absence of ED and on adherence to the National Institute of Health's definition of ED. These items focus on erectile function and intercourse satisfaction. The items are rated on a scale from 1-5 (e.g., 1=Very low to 5=Very high; 1=Almost never/never to 5=Almost always/always; 1=Extremely difficult to 5=Not difficult). The IIEF-5 score is the sum of questions 1 to 5 (Scores range from 5-25). ED was classified into five severity levels, ranging from none (22-25) through severe (5-7).
Development of International prostate symptom score (IPSS) compared to baseline | Preoperatively (Baseline), 6 weeks, 3 months and 6 months postoperatively.
  The International prostate symptom score (IPSS) questionnaire has seven questions, which are used to evaluate storage and voiding symptoms. The patient is given ﬁve options for the ﬁrst seven questions and each option indicates severity of that symptom. The total score ranges from 0 to 35 and Lower Urinary Tract Symptoms (LUTS) are classiﬁed as mild to severe depending on the total score. Patients having a total score ≤7 are classiﬁed as having mild symptoms, scores from 8 to 19 are classiﬁed as moderate symptoms, and symptom scores ≥20 are classiﬁed as severe symptoms.
Comparison of Prostate Specific Antigen (PSA) at screening and 6 weeks after surgery. | at screening and 6 weeks after surgery.
  PSA response will be measured as the change of serum PSA in ng/mL between preoperative / screening examination and at follow-up 6 weeks after surgery

OTHER OUTCOMES:
Assessment of the intraoperative handling of the Symmcora® Long bidirectional | after inclusion of the last patient
  Handling of the suture is assessed for every participating surgeon once after inclusion of the last patient. Handling is measured in 16 dimensions + overall impression with five evaluation levels (excellent, very good, good, satisfied, poor)
Assessment of the intraoperative handling of the Symmcora® Mid Unidirectional | after inclusion of the last patient
  Handling of the suture is assessed for every participating surgeon once after inclusion of the last patient. Handling is measured in 13 dimensions + overall impression with five evaluation levels (excellent, very good, good, satisfied, poor)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Miguel Sánchez Encinas, Dr., Principal Investigator — Hospital Universitario Rey Juan Carlos
Locations (2):
- Spain (2):
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid